CLINICAL TRIAL: NCT06019117
Title: Effectiveness of a Probiotic K10 in Managing Health Outcomes in Parkinson's Disease and in Early Stage (Mild Cognitive Impairment to Mild Dementia) and Alzheimer's Disease
Brief Title: Effectiveness of Probiotic K10 in Managing Health Outcomes in Parkinson and Alzheimer Disease
Acronym: Probiótico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deivis de Oliveira guimaraes (Network)
Responsible Party: Sponsor-Investigator, Deivis de Oliveira guimaraes, Director of Research, Gon1 Gestao de Projetos
Organization: Gon1 Gestao de Projetos (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023001
Record Dates: First submitted 2023-08-17; First posted 2023-08-31 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease; Alzheimer Disease
Keywords: Probiotic; Alzheimer; Parkinson; Neurological desease
MeSH Terms: conditions — Parkinson Disease; Alzheimer Disease | interventions — Flour

STUDY DESIGN:
Intervention Model Description: Single-centre, double-blind, placebo-controlled randomized clinical trial (RCT), Interventional Model: Parallel Assignment, phase III study.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 - volunteers with parkinson's disease (Active Comparator): 26 patients in this arm. in this arm will receive the probiotic K10 (30.000.000 CFU/day).
  Interventions: Dietary Supplement: Probiotic K10
- Arm 2 - volunteers with parkinson's disease (Placebo Comparator): 26 patients in this arm. In this arm will receive the controlled placebo.
  Interventions: Drug: Placebo
- Arm 3- volunteers with alzheimer's disease (Active Comparator): 26 patients in this arm. in this arm will receive the probiotic K10 (30.000.000 CFU/day).
  Interventions: Dietary Supplement: Probiotic K10
- Arm 4- volunteers with alzheimer's disease (Placebo Comparator): 26 patients in this arm. In this arm will receive the controlled placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic K10 — clinical trial using 90 days of probiotic K10
  Other Names: Mix probiotic; Neurobiotic
  Arms: Arm 1 - volunteers with parkinson's disease; Arm 3- volunteers with alzheimer's disease
Drug: Placebo — clinical trial using 90 days of placebo controlled
  Other Names: flour
  Arms: Arm 2 - volunteers with parkinson's disease; Arm 4- volunteers with alzheimer's disease

SUMMARY:
Evaluation of the effects of the K10 probiotic mix in patients with degenerative neurological diseases (Parkinson and Alzheimer's) with a focus on cognitive, motor and psychiatric neurological evaluation.

Single-centre, double-blind, placebo-controlled randomized clinical trial (RCT), Interventional Model: Parallel Assignment, phase III study. Two groups will be composed, with two arms each, 1 group composed of patients with Parkinson's and 1 group with patients with Alzheimer's, 52 patients in each group. The first arm of each group will receive placebo and the other arm of each group will receive the mix K10.

In this study, researchers will conduct a randomized, placebo-controlled, phase III trial of a probiotic preparation (Probiotic K10) to evaluate its use as a viable treatment option for neurodegenerative disorders, including Parkinson's disease (PD) and Alzheimer's disease. of Alzheimer (AD). This formulation has been previously demonstrated to improve cognitive function, systemic inflammation, systemic oxidative stress in Alzheimer's patients. The main objective of this study is to compare its effect with placebo on cognitive status in individuals with AD and PD, the UPDRS total score in people with early PD and quality of life, and the measurement of caregiver burden in AD and PD. Participants will be randomly assigned to receive a placebo (an inactive substance) and a K10 probiotic (dose 30.000.000 CFU/day). They will be evaluated at baseline, 45 days and 90 days.

DETAILED DESCRIPTION:
Change in urinary cortisol dosage Determination of cortisol levels can be used as an indirect measurement of emotional stress. Reduced levels of this hormone are related to reduced cardiovascular risk and reduced inflammatory damage.

Baseline to T90 or the time of sufficient disability to study closure.

All measurements will be taken at time zero (start of the survey), the next measurement in 45 days and the last measurement in 90 days. We will use the comparison of the data collected from each individual at time zero in comparison with their own results collected at the next times, using biostatistics to compare the results and, at the end of the primary result, we will perform the simple tabulation to count the values of each analyzed variable.

Differences between measures of central tendency with pr < 0.05 will be considered statistically significant. When the central tendency values present a normal distribution in the statistical test, a parametric test will be used. In the case of comparison of 2 means, Student's t test will be used, for paired or independent samples. When the comparison includes more than 2 means, analysis of variance (ANOVA) will be used for 1 way (a single factor, e.g. treatment time) or 2 ways (two factors, for example treatment time and control group x treated group ).

After verifying a significant difference in ANOVA, a post hoc protected t-test will then be applied to detect at which points in the analysis there are pairs with significant differences. When the analysis of the distribution (frequency) of the data shows a distribution that is not compatible with the Gaussian distribution, a corresponding non-parametric test will be used. Contingency tables 2 x 2 will also be used for later calculation of risk factors and to determine the significance through the X2 test.

The software to be used will be Prism from Graphpad v. 9

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for individuals with Parkinson's. Ages eligible to participate in the study: 18 years or older Accept healthy volunteers: No. Gender Eligibility for Study: All genders

Inclusion criteria:

* Presence of all 3 cardinal features of Parkinson's disease (tooth tremor, bradykinesia, and rigidity). Clinical signs must be asymmetrical.
* Diagnosis of Parkinson's disease within 5 years of the Screening Visit.
* Age 18 years or older.
* Women must not be of childbearing potential or must use an approved form of contraception during the trial period.

Eligibility Criteria for Individuals with Alzheimer's. Eligible ages to participate in the study: 60 -85 years Accept healthy volunteers: No. Gender Eligibility for Study: All genders

Inclusion criteria:

* Men or women between the ages of 60 and 85
* Diagnosis of probable Alzheimer's disease
* Portuguese-speaking, English-speaking; Spanish-speaking if the individual site allows
* Study partner or caregiver to ensure compliance
* Mini-Mental State Exam score at screening visit greater than 14
* Stable medical condition for 3 months prior to screening, with no significant abnormal liver, kidney, or blood studies.
* Able to take oral medications
* Modified Hachinski Ischemic Index less than or equal to 4
* CT or MRI from the onset of memory impairment, demonstrating the absence of a clinically significant focal lesion
* Physically acceptable for this study, as confirmed by medical history, physical examination, neurological examination, and clinical testing

Exclusion Criteria:

Parkinson's Exclusion Criteria:

* Parkinsonism due to drugs including neuroleptics, alpha-methyldopa, reserpine, metoclopramide, valproic acid.
* Use of antioxidants (such as selegiline, rasagiline, vitamins E and C), additional supplemental vitamins or minerals, regular use of neuroleptics, chloramphenicol, valproic acid, warfarin.
* Other parkinsonian disorders.
* Modified Hoehn and Yahr score of 3 or more on Screening Visit or Baseline Visit.
* UPDRS tremor score of 3 or greater at Screening Visit or Baseline Visit.
* History of symptomatic stroke.
* Sufficient deficiency to require changes in dopaminergic medication treatment during follow-up compared to baseline treatment schedule.
* Other severe and uncompensated illnesses, including severe psychiatric illnesses.
* Patients with active cardiovascular, restrictive peripheral vascular, or cerebrovascular disease in the past year.
* Unstable dose of active CNS therapies.
* Use of appetite suppressants within 60 days of the Baseline Visit.
* History of active epilepsy within the past 5 years.
* Participation in other drug studies or use of other investigational drugs within 30 days prior to the Screening Visit.
* History of electroconvulsive therapy.
* History of any brain surgery for Parkinson's disease.
* History of structural brain disease, such as previous trauma causing damage detected on a CT scan or MRI, hydrocephalus, or previous brain neoplasms.

Alzheimer's Exclusion Criteria:

* Significant neurological disease such as Parkinson's disease, stroke, brain tumor, multiple sclerosis, or seizure disorder
* Major depression treated in the past 12 months, major mental illness such as schizophrenia, or recent (in past 12 months) alcohol or substance abuse
* History of invasive cancer within the past two years (excluding non-melanoma skin cancer)
* Use of any investigational agents within 30 days prior to screening
* Major surgery within 8 weeks prior to the Baseline Visit
* Uncontrolled cardiac conditions or severe unstable medical illnesses
* Antiretroviral therapy for human immunodeficiency virus (HIV)
* Conditions that will contribute to oxidative stress: current cigarette or cigar smokers (within past month), diabetics on insulin or poorly controlled on oral hypoglycemics
* Blindness, deafness, language difficulties or any other disability which may prevent the participant from participating or cooperating in the protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Parkinson under 18 years. Alzheimer between 60 and 85 years
Enrollment: 104 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2024-01-07 (Actual)

PRIMARY OUTCOMES:
Change in MDS-Unified (PD) | 1st, 45 and 90 days
  scale (MDS- UPDRS) the sum of parts I, II and III ranges from 0 to 176. The MDS-UPDRS score has three components, each consisting of questions with 0-4 point scale. Part I assesses mentation, behavior, and mood; Part II assesses activities of daily; and Part III assesses motor abilities. Where 0 represents the absence of impairment and 4 represents the highest degree of impairment.
Change in quality of life scale (PD) | 1st, 45 and 90 days
  Questionnaire (PDQ-39) that will evaluate their health and overall quality of life. The total of 39 aspects of quality of life, maximum score is 132. Each aspect is rated on scale of 0 (best outcome) to 4 (worst outcome). A higher score or increased score compared to a previous visit indicates a lowered quality of life.
Changes in anxiety levels (PD&AD) | 1st, 45 and 90 days
  Changes in anxiety levels, mood improvement and caregiver burden will be determined by applying the Neuropsychiatric Questionnaire (NPI-Q)
Changes in cognitive status measured by brief battery (AD) | 1st, 45 and 90 days
  Mini Mental State Examination (MMSE): maximum score 30 points. Higher values indicate greater cognitive performance.
Change in Quality of Life (QOL) (AD) | 1st, 45 and 90 days
  13-item QOL-AD scale (total score range 13-52; higher scores indicate better QOL). The QOL-AD scale uses 1-4 (poor, fair, good, or excellent) to rate a variety of life domains, including the patient's physical health, mood, relationships, activities, and ability to complete tasks.

SECONDARY OUTCOMES:
Change in cortisol dosage (Parkinson's and Alzheimer's group) | 1st, 45 and 90 days
  Determination of cortisol levels can be used as an indirect measurement of emotional stress. Reduced levels of this hormone are related to reduced cardiovascular risk and reduced inflammatory damage.

CONTACTS AND LOCATIONS:
Overall Officials: Alyne M Ton, post-doc, Principal Investigator — Gon1 Gestora de Projetos; Sarha A L Queiroz, PhD, Principal Investigator — Gon1 Gestora de Projetos; Deivis O Guimaraes, Mba, Study Director — Gon1 Gestora de Projetos
Locations (1):
- Gon1 gestora de Projetos, Vitória, Espírito Santo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We can share all data regarding data collection, preserving the personal data of volunteers and as long as the request does not go beyond the limits of confidentiality, integrity and ethics.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: They will be available after data collection and analysis, and will be abble for 1 year after the trial end.
Access Criteria: will be available upon request and for exclusive access to scientists, governmental and scientific organizations.
URL: https://gon1.com.br/DP-DA.html

REFERENCES:
- [Background] Mazloom Z, Yousefinejad A, Dabbaghmanesh MH. Effect of probiotics on lipid profile, glycemic control, insulin action, oxidative stress, and inflammatory markers in patients with type 2 diabetes: a clinical trial. Iran J Med Sci. 2013 Mar;38(1):38-43. PMID 23645956
- [Background] Liu Z, Li T, Li P, Wei N, Zhao Z, Liang H, Ji X, Chen W, Xue M, Wei J. The Ambiguous Relationship of Oxidative Stress, Tau Hyperphosphorylation, and Autophagy Dysfunction in Alzheimer's Disease. Oxid Med Cell Longev. 2015;2015:352723. doi: 10.1155/2015/352723. Epub 2015 Jun 15. PMID 26171115
- [Background] Mishra V, Shah C, Mokashe N, Chavan R, Yadav H, Prajapati J. Probiotics as potential antioxidants: a systematic review. J Agric Food Chem. 2015 Apr 15;63(14):3615-26. doi: 10.1021/jf506326t. Epub 2015 Apr 6. PMID 25808285
- [Background] Licker V, Kovari E, Hochstrasser DF, Burkhard PR. Proteomics in human Parkinson's disease research. J Proteomics. 2009 Nov 2;73(1):10-29. doi: 10.1016/j.jprot.2009.07.007. Epub 2009 Jul 24. PMID 19632367
- [Background] Alexander GE, Crutcher MD, DeLong MR. Basal ganglia-thalamocortical circuits: parallel substrates for motor, oculomotor, "prefrontal" and "limbic" functions. Prog Brain Res. 1990;85:119-46. PMID 2094891
- [Background] Obeso JA, Rodriguez-Oroz MC, Chana P, Lera G, Rodriguez M, Olanow CW. The evolution and origin of motor complications in Parkinson's disease. Neurology. 2000;55(11 Suppl 4):S13-20; discussion S21-3. PMID 11147505
- [Background] Sood B, Patel P, Keenaghan M. Coenzyme Q10. 2024 Jan 30. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK531491/ PMID 30285386
- [Background] Arenas-Jal M, Sune-Negre JM, Garcia-Montoya E. Coenzyme Q10 supplementation: Efficacy, safety, and formulation challenges. Compr Rev Food Sci Food Saf. 2020 Mar;19(2):574-594. doi: 10.1111/1541-4337.12539. Epub 2020 Feb 19. PMID 33325173
- [Background] Garrido-Maraver J, Cordero MD, Oropesa-Avila M, Vega AF, de la Mata M, Pavon AD, Alcocer-Gomez E, Calero CP, Paz MV, Alanis M, de Lavera I, Cotan D, Sanchez-Alcazar JA. Clinical applications of coenzyme Q10. Front Biosci (Landmark Ed). 2014 Jan 1;19(4):619-33. doi: 10.2741/4231. PMID 24389208
- [Result] Valentini L, Pinto A, Bourdel-Marchasson I, Ostan R, Brigidi P, Turroni S, Hrelia S, Hrelia P, Bereswill S, Fischer A, Leoncini E, Malaguti M, Blanc-Bisson C, Durrieu J, Spazzafumo L, Buccolini F, Pryen F, Donini LM, Franceschi C, Lochs H. Impact of personalized diet and probiotic supplementation on inflammation, nutritional parameters and intestinal microbiota - The "RISTOMED project": Randomized controlled trial in healthy older people. Clin Nutr. 2015 Aug;34(4):593-602. doi: 10.1016/j.clnu.2014.09.023. Epub 2014 Oct 8. PMID 25453395
- [Result] Padurariu M, Ciobica A, Lefter R, Serban IL, Stefanescu C, Chirita R. The oxidative stress hypothesis in Alzheimer's disease. Psychiatr Danub. 2013 Dec;25(4):401-9. PMID 24247053
- [Result] Blum D, Torch S, Lambeng N, Nissou M, Benabid AL, Sadoul R, Verna JM. Molecular pathways involved in the neurotoxicity of 6-OHDA, dopamine and MPTP: contribution to the apoptotic theory in Parkinson's disease. Prog Neurobiol. 2001 Oct;65(2):135-72. doi: 10.1016/s0301-0082(01)00003-x. PMID 11403877